CLINICAL TRIAL: NCT05336695
Title: Assess the Brain Levels of Fibrin in Alzheimer's Disease and Its Related Dementias Subjects Using 64Cu-FBP8 PET
Brief Title: Assess Fibrin in Brains With AD/ADRD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ciprian Catana, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019P002911; 3R01HL109448-07S1 (NIH)
Record Dates: First submitted 2022-04-06; First posted 2022-04-20 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer Disease; Dementia of Alzheimer Type
Keywords: Alzheimer Disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Positron-Emission Tomography; Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: All subjects will receive the same injection of 64Cu-FBP8 and undergo PET/MR imaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Cognitively Normal Subjects and ADRD subjects (Experimental): Cognitively Normal Subjects and ADRD subjects
  Interventions: Diagnostic Test: PET/MR Imaging; Drug: 64Cu-FBP8

INTERVENTIONS:
Diagnostic Test: PET/MR Imaging — PET/MRI Scan with [64Cu]FBP8 as directed by protocol
  Other Names: Positron Emission Tomography/Magnetic Resonance Imaging
Drug: 64Cu-FBP8 — Will be administered by intravenous injection by bolus by a qualified nuclear medicine technician at the Martinos Center
  Other Names: Positron Emission Tomography dye

SUMMARY:
The goal of this project is to quantify brain fibrin content using 64Cu-FBP8-PET in the brains of subjects ranging from cognitively normal to clinically diagnosed with ADRD to evaluate potential regional differences.

DETAILED DESCRIPTION:
While there are many potential therapeutics being evaluated for Alzheimer's disease and related dementias (ADRD), there is currently no known cure for ADRD and its origin and pathophysiology are still not well understood. However, the association of fibrin with ADRD is becoming increasingly clearer. Up to now it was not possible to quantify brain fibrin in vivo to better elucidate its role in ADRD, but recently, 64Cu-FBP8 was proposed as a tool to detect thrombus anywhere in the body. This unique tool will allow us to non-invasively assess brain fibrin levels in at-risk and ADRD subjects.

The goal of this project is to use 64Cu-FBP8-PET in the brains of subjects ranging from cognitively normal to clinically diagnosed with ADRD to assess fibrin levels. It is expected that about 30 people will take part in this research study. 64Cu-FBP8-PET is not currently approved by the U.S. Food and Drug Administration (FDA).

ELIGIBILITY:
Inclusion Criteria:

* Age between 55 and 90 years
* Ability to provide informed consent
* Specific to healthy volunteers: no history of ADRD
* Specific to ADRD subjects: clinical diagnosis of AD - either amnestic or atypical, clinical severity ranging from MCI to moderate dementia (CDR 0.5-2.0), MMSE score greater than or equal to 15 and/or MOCA greater than or equal to 12
* Specific to BAnD subjects: referred through the Brain Aging and Dementia (BAnD) research registry

Exclusion Criteria:

* MR contraindications such as: electrical implants such as cardiac pacemakers or perfusion pumps; ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants, ferromagnetic objects such as jewelry or metal clips in clothing
* Preexisting medical conditions including a likelihood of developing seizures or claustrophobic reactions, and any greater than normal potential for cardiac arrest
* Subjects whose estimated glomerular filtration rate (eGFR) < 60 mL/min will be excluded from receiving the gadolinium-based contrast agent
* Research-related radiation exposure exceeding current Massachusetts General Hospital (MGH) Radiology Department guidelines (i.e. 50 millisievert in the prior 12 months)
* 3. In line with published MGH IRB guidelines for pregnancy must be ruled out by urine ß-HCG if answers to screening questions suggest that pregnancy is possible and if female participants are premenopausal and of child-bearing age. Subjects will not be able to enroll if they are breastfeeding.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2026-09-28 (Estimated); Study Completion 2026-09-28 (Estimated)

PRIMARY OUTCOMES:
Concentration of fibrin in the brains of ADRD subjects and healthy controls | baseline
  64Cu-FBP8-PET will be used to quantify brain fibrin content in the brains of ADRD subjects and healthy controls to evaluate potential regional differences.

CONTACTS AND LOCATIONS:
Overall Officials: Ciprian Catana, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States